CLINICAL TRIAL: NCT00750256
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of GSK1278863A in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK1278863A in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PHX111427
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Anaemia
Keywords: tolerability; Safety; pharmacokinetics
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohorts (Experimental): This study will be a single-blind, randomized, placebo-controlled, dose-rising, single dose, parallel group study with 6 proposed Cohorts from 2mg to 450mg.
  Interventions: Drug: GSK1278863A

INTERVENTIONS:
Drug: GSK1278863A — GSK1278863A planned doses from 2mg to 450mg which may change based on safety or PK from previous cohorts.

SUMMARY:
A first-time in human study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK1278863A in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking (within 40 days of screening), adult males and females between 18 and 55 years of age, inclusive
* Female subjects are eligible for participation in the study if they are of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant);
* Male subjects agree to use contraception methods
* Body weight > or = 50 kg; BMI: 19-31 kg/m2, inclusive
* Subject has a QTc <450 msec or <480 msec if associated with bundle branch block
* Subject is willing and able to provide written informed consent

Exclusion Criteria:

* MCV value outside the reference range at screening
* Hemoglobin value at screening is: male subjects or post-menopausal females > 15.5 g/dL; female subjects > 14.5 g/dL
* TIBC, serum iron and serum ferritin values are outside the reference range at screening
* Calculated creatinine clearance < 60 ml/min
* Clinically significant abnormal CPK determined by the investigator and medical monitor
* AST, ALT and direct bilirubin are greater than upper limit of reference range at screening
* Subjects are unwilling or inability to follow the procedures and lifestyle and/or dietary restrictions outlined in the protocol
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures or compromise subject safety
* Subject currently exposures to more than four new chemical entities within 12 months prior to the first dosing day
* Use of other prescription or non-prescription drugs, vitamins, herbal and dietary supplements, within 7 days prior to the first dose of study medication
* Subject has a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Subject has a history of GI ulceration or gastrointestinal bleeding
* Subject has a history of peptic ulcer disease
* Subject has a history of malignancy tumor; non-melanoma skin cancer that has been definitely removed is allowed
* Treatment with an investigational drug within 30 days preceding the first dose of study medication
* Subjects with a history of drug abuse
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening
* Positive urine drug screen (UDS) at screening
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result or positive HIV result within 3 months of screening
* Donation of blood in excess of 500 mL within 56 days prior to first dose of study medication
* Subject has a history of regular use of tobacco- or nicotine containing products
* History of sensitivity to heparin, heparin-induced thrombocytopenia or sensitivity to any of the study medications or components thereof

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-07-07 (Actual); Primary Completion 2008-12-12 (Actual); Study Completion 2008-12-12 (Actual)

PRIMARY OUTCOMES:
GSK1278863A safety endpoints: adverse events reporting, clinical safety laboratory tests (hematology, chemistry, urinalysis,and fecal occult blood), vital signs, 12-lead ECG, dual-lead cardiac monitoring. | 1 Day

SECONDARY OUTCOMES:
Blood and urine levels of GSK1278863A | 2 Days
Effect of GSK1278863A on hematological markers | 2 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States

REFERENCES:
- See also: Results for study PHX111427 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/PHX111427?search=study&search_terms=PHX111427#rs